CLINICAL TRIAL: NCT01224158
Title: Efficacy of an Experimental Toothbrush on the Treatment and Prevention of Gingivitis
Brief Title: Study of an Experimental Toothbrush for Treatment and Prevention of Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: TBRGBP0016
Record Dates: First submitted 2010-10-15; First posted 2010-10-19 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Dental Devices, Home Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- PR-009577 Toothbrush (Experimental): Experimental Power Toothbrush
  Interventions: Device: Experimental Power Toothbrush
- PR-000172 Toothbrush (Active Comparator): Flat trimmed Manual Toothbrush
  Interventions: Device: Flat trimmed Manual Toothbrush

INTERVENTIONS:
Device: Experimental Power Toothbrush — Following a placebo mouthwash phase, Subjects will be asked to brush their teeth (twice per day with the experimental toothbrush and toothpaste provided) moving to the next quadrant of the mouth at 30-second intervals.
  Other Names: Not yet marketed
  Arms: PR-009577 Toothbrush
Device: Flat trimmed Manual Toothbrush — Following a placebo mouthwash phase, Subjects will be asked to brush their teeth (twice per day using the toothbrush and toothpaste provided) in their usual manner.
  Other Names: Reach®
  Arms: PR-000172 Toothbrush

SUMMARY:
This study is 6 weeks long with 6 visits to a clinical site. People participating in this study will be asked to brush their teeth two times a day with a provided toothbrush. For one of those six weeks people will be asked to rinse with a mouthwash. During that time, people will use the mouthwash two times a day and will not be allowed to brush their teeth at all. The mouth, teeth, tongue and gums will be looked at by a dentist. At each visit, people will rinse with a pink liquid that will dye their mouths pink. The dye is temporary and will go away by the end of the day. They may also be asked to complete a short questionnaire about their experience.

DETAILED DESCRIPTION:
This is a 42-day, randomized, observer-blind, parallel group, single-center clinical trial. Generally healthy adults will be recruited from a database of known plaque formers. A sufficient number of subjects meeting the necessary inclusion/exclusion criteria will be enrolled into two groups, so that 140 subjects (70 per treatment group) would reasonably be expected to complete the study.

The study will have a pre-experimental phase, which will last 2 weeks followed by an experimental phase that is 4 weeks in duration. At the start of the pre-experimental phase (Day 0), subjects will undergo an initial oral exam, during which gingivitis and pre-brushing plaque evaluations will be performed. Supragingival plaque levels will be assessed on all scorable teeth according to the Rustogi Modified Navy Plaque Index (RMNPI) and gingivitis will be scored according to the Modified Gingival Index (MGI). Subjects with a whole mouth mean plaque level > 0.60 and a whole mouth mean MGI ≥ 1.75 will then brush their teeth with their assigned toothbrush using American Dental Association (ADA) Accepted fluoride toothpaste. They will be provided with written and verbal instructions to use their toothbrush twice a day, for the next 7 days (Normalization period), allowing the participants to get familiar with the assigned test product. During the second visit (Day 7), the subjects will return the products to the clinical site, and start the experimental gingivitis phase, during which they will only be allowed to use a placebo rinse (W002194-0221P) as means of oral hygiene. The objective of the experimental gingivitis phase is to standardize the levels of plaque and gingivitis in both groups.

At visit 3 (Day 14), subjects will undergo a second gingivitis and pre-brushing plaque evaluation and receive their assigned brush, instructions and diary. They will brush with their assigned toothbrush for two weeks (14 days), using an ADA accepted fluoride toothpaste. During the fourth visit (Day 28), the subjects will return to the site and undergo a third gingivitis and post-brushing plaque evaluation. At the last visit (Day 42), the study participants will undergo final gingivitis and post-brushing plaque evaluations and return all used products.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age and in good general and oral health.
* Evidence of a personally signed and dated informed consent document indicating the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial.
* Willingness to use the assigned products according to instructions, availability for appointments and likelihood of completing the clinical trial.
* Good general and oral health with manual dexterity.
* Willingness to refrain from all oral hygiene procedures within 18-24 hours prior to the study visit.
* A minimum of twenty scorable teeth with at least one scorable molar in each quadrant.
* A whole-mouth mean plaque level greater than 0.60 at Day 0.
* Whole-mouth-mean gingivitis level greater than or equal to 1.75 at Day 0.
* Absence of orthodontic bands, appliances, bridges, numerous crowns, extensive large restorations, excessive caries, removable orthodontic appliances or partial dentures.
* Absence of significant oral soft tissue pathology, excluding gingivitis, based on the visual oral examination and at the discretion of the examiner.
* Adequate oral hygiene (i.e., brush teeth daily and exhibit no signs of oral neglect).
* Absence of moderate/advanced periodontitis.
* Absence of extensive supragingival calculus.
* Absence of ulcerations on lips and oral mucosa.

Exclusion Criteria:

* Currently taking steroids, antibiotic medication or any other medication within the previous month that may interfere with the efficacy evaluations.
* Those requiring antibiotic premedication prior to dental treatment.
* Participation in a dental clinical trial involving oral care products currently or within the past 28 days.
* Dental prophylaxis within one week prior to enrollment into the study.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.
* Physical limitations or restrictions that might preclude use of normal oral hygiene procedures (i.e., toothbrushing, etc.).
* Self-reported pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2010-09-13 (Actual); Primary Completion 2010-10-29 (Actual); Study Completion 2010-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Araujo, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (1):
- BioSci Research America, Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Manual Toothbrush (PR-000172): Following a placebo rinse phase of 7 days, participants brushed their teeth (twice per day using the PR-000172 toothbrush and toothpaste provided) in their usual manner up to Day 42.
- Power Toothbrush (PR-009577): Following a placebo rinse phase for 7 days, Participants brushed their teeth (twice per day with the experimental toothbrush PR-009577 and toothpaste provided) up to Day 42.
Period: Overall Study
Arm/Group | Manual Toothbrush (PR-000172) | Power Toothbrush (PR-009577)
Started | 76 | 77
Completed | 75 | 77
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Toothbrush (PR-000172) | Power Toothbrush (PR-009577) | Total
Number analyzed (Participants) | 76 | 77 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (10.21) | 32.9 (9.61) | 32.7 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 46 | 88
  Male | 34 | 31 | 65
Region of Enrollment [Count of Participants; unit: Participants]
  United States: USA | 76 | 77 | 153

OUTCOME MEASURES:

1. Primary Outcome: Whole-mouth Mean Modified Gingival Index (MGI) Score at Day 42
Description: Gingivitis was assessed by the Modified Gingival Index on the buccal and lingual marginal gingiva and interdental papillae of all scorable teeth by the dental examiner using following scale score range from 0 to 4, where 0 - Normal (absence of inflammation); 1 - Mild inflammation (slight change in color, little change in texture) of any portion of the gingival unit; 2 - Mild inflammation of the entire gingival unit; 3 - Moderate inflammation (moderate glazing, redness, edema, and/or hypertrophy) of the gingival unit; 4 - Severe inflammation (marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration) of the gingival unit.
Time Frame: Day 42
Population: Full Analysis Set (FAS), included all randomized participants who have MGI at Day 0 and at least one MGI value on Day 28 or Day 42.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Manual Toothbrush (PR-000172) | Power Toothbrush (PR-009577)
Number analyzed (Participants) | 75 | 77
Unit on a scale | 1.880 (0.1223) | 1.770 (0.1443)

2. Secondary Outcome: Whole-mouth Mean Modified Gingival Index (MGI) Score at Day 28
Description: Gingivitis was assessed by the Modified Gingival Index on the buccal and lingual marginal gingiva and interdental papillae of all scorable teeth by the dental examiner using following scale with score range from 0 to 4, where 0 - Normal (absence of inflammation); 1 - Mild inflammation (slight change in color, little change in texture) of any portion of the gingival unit; 2 - Mild inflammation of the entire gingival unit; 3 - Moderate inflammation (moderate glazing, redness, edema, and/or hypertrophy) of the gingival unit; 4 - Severe inflammation (marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration) of the gingival unit.
Time Frame: Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Manual Toothbrush (PR-000172) | Power Toothbrush (PR-009577)
Number analyzed (Participants) | 75 | 77
Unit on a scale | 1.957 (0.1225) | 1.868 (0.1287)

3. Secondary Outcome: Whole-mouth Mean Rustogi Modified Navy Plaque Index (RMNPI) Score at Day 42
Description: Supra-gingival plaque was assessed on the facial and lingual surfaces of the teeth (7-7 each arch) using the RMNPI. The facial and lingual surfaces were divided into nine unequal segments, as follows, for a total of 18 sites per tooth: A-C along the gingival margin; D and F (inter-proximal zones) directly above A-C; G-H across the middle of the tooth and I covers the incisal area. Plaque was assigned on one of the following score: 0 represents no dental plaque and 1 represents plaque present in the measured segment of the tooth. Mean RMNPI overall was calculated for each participant as the total score for all tooth sites assessed divided by the total number of tooth sites assessed.
Time Frame: Day 42
Population: FAS included all randomized participants who have MGI at Day 0 and at least one MGI value on Day 28 or Day 42.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Manual Toothbrush (PR-000172) | Power Toothbrush (PR-009577)
Number analyzed (Participants) | 75 | 77
Units on a scale | 0.146 (0.0710) | 0.131 (0.0633)

4. Secondary Outcome: Whole-Mouth Mean Rustogi Modified Navy Plaque Index (RMNPI) Score at Day 28
Description: as for outcome 3
Time Frame: Day 28
Population: FAS included all randomized participants who have MGI at Day 0 and at least one MGI value on Day 28 or Day 42.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Manual Toothbrush (PR-000172) | Power Toothbrush (PR-009577)
Number analyzed (Participants) | 75 | 77
Units on a scale | 0.164 (0.0755) | 0.148 (0.0762)

5. Secondary Outcome: Hard-to-reach Mean Rustogi Modified Navy Plaque Index (RMNPI) at Day 28 and 42
Description: Hard-to-reach mean score is defined as mean of scores over following areas combined; a) Gingival margin (Sites A - C); b) Distal Molars (F for teeth 2, 15, 18, and 31 or the most posterior molar in that quadrant); c) Lingual of the mandibular incisors (Teeth 23-26, lingual); d) Interproximal (Sites D and F); e) Mandibular posterior lingual (Teeth 18-21, 28-31, lingual). Supra-gingival plaque was assessed on facial and lingual surfaces of teeth (7-7 each arch) using the RMNPI. The facial and lingual surfaces were divided into nine unequal segments, as follows, for a total of 18 sites per tooth: A-C along gingival margin; D and F (inter-proximal zones) directly above A-C; G-H across middle of tooth and I covers incisal area. Plaque was disclosed on a scale (0 indicates no dental plaque to 1 indicates dental plaque), Mean RPI overall was calculated for each participant as total score for all tooth sites assessed divided by total number of tooth sites assessed.
Time Frame: Day 28 and 42
Population: FAS included all randomized participants who have MGI at Day 0 and at least one MGI value on Day 28 or Day 42.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Manual Toothbrush (PR-000172) | Power Toothbrush (PR-009577)
Number analyzed (Participants) | 75 | 77
Units on a scale
  Day 28 | 0.232 (0.1066) | 0.209 (0.1067)
  Day 42 | 0.208 (0.0993) | 0.186 (0.0905)

6. Secondary Outcome: Mean Rustogi Modified Navy Plaque Index (RMNPI) at Day 28 and 42 for Each Hard-to-reach Area
Description: Hard-to-reach mean score is defined as mean of scores over following areas separately d; a) Gingival margin (Sites A - C); b) Distal Molars (F for teeth 2, 15, 18, and 31 or the most posterior molar in that quadrant); c) Lingual of the mandibular incisors (Teeth 23-26, lingual); d) Interproximal (Sites D and F); e) Mandibular posterior lingual (Teeth 18-21, 28-31, lingual). Supra-gingival plaque was assessed on facial and lingual surfaces of teeth (7-7 each arch) using the RMNPI. The facial and lingual surfaces were divided into nine unequal segments, as follows, for a total of 18 sites per tooth: A-C along gingival margin; D and F (inter-proximal zones) directly above A-C; G-H across middle of tooth and I covers incisal area. Plaque on each area was assigned one of the following score: on a scale (0 indicates no dental plaque and 1 indicates plaque present in the measured segment of the tooth).
Time Frame: Day 28 and 42
Population: FAS included all randomized participants who have MGI at Day 0 and at least one MGI value on Day 28 or Day 42.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Manual Toothbrush (PR-000172) | Power Toothbrush (PR-009577)
Number analyzed (Participants) | 75 | 77
Units on a scale
  Gingival Margin: Day 28 | 0.298 (0.1172) | 0.271 (0.1169)
  Gingival Margin: Day 42 | 0.273 (0.1181) | 0.246 (0.0992)
  Distal Molars: Day 28 | 0.413 (0.2599) | 0.399 (0.2175)
  Distal Molars: Day 42 | 0.352 (0.2172) | 0.339 (0.2284)
  Lingual of the Mandibular Incisors: Day 28 | 0.190 (0.2501) | 0.149 (0.2430)
  Lingual of the Mandibular Incisors: Day 42 | 0.152 (0.1892) | 0.119 (0.2035)
  Interproximal: Day 28 | 0.195 (0.1173) | 0.169 (0.1122)
  Interproximal: Day 42 | 0.171 (0.1047) | 0.148 (0.1054)
  Mandibular Posterior Lingual: Day 28 | 0.368 (0.1808) | 0.372 (0.1888)
  Mandibular Posterior Lingual: Day 42 | 0.351 (0.1789) | 0.336 (0.1473)

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Description: Safety Analysis Set includes all participants who use clinical trial test product and have any follow-up information.
Arm/Group | Manual Toothbrush (PR-000172) | Power Toothbrush (PR-009577)
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/77
Other Adverse Events (participants affected / at risk) | 0/76 | 0/77

LIMITATIONS AND CAVEATS:
No study limitations were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.